CLINICAL TRIAL: NCT07291752
Title: The Risk of Second Primary Gastrointestinal Malignancies Following Primary Gastrointestinal Carcinoid Tumors: a SEER Based Study 2000-2022
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Other Study IDs: A276
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Carcinoid Tumor; Second Primary Malignant Neoplasm
Keywords: SEER; Carcinoid; malignancy
MeSH Terms: conditions — Carcinoid Tumor; Neoplasms, Second Primary; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carcinoid tumors are rare neuroendocrine tumors with slowly progressive course. Carcinoid tumors are the most common gastrointestinal (GI) neuroendocrine tumors. The most common sites of GI carcinoids are small intestine accounting for 45%, rectum (20%), appendix (17%), colon (11%), and stomach (7%). Some studies reported an association between neuroendocrine tumors and multiple malignancies. However, the presence of neuroendocrine tumors combined with multiple primary GI tumors is considered an exotic event in the literature with only few case studies and case series. So the aim of this study is to assess the risk of GI malignancies following primary GI carcinoids.

DETAILED DESCRIPTION:
Carcinoid tumors are rare neuroendocrine tumors with slowly progressive course. Carcinoid tumors are the most common gastrointestinal (GI) neuroendocrine tumors. The most common sites of GI carcinoids are small intestine accounting for 45%, rectum (20%), appendix (17%), colon (11%), and stomach (7%). Some studies reported an association between neuroendocrine tumors and multiple malignancies. However, the presence of neuroendocrine tumors combined with multiple primary GI tumors is considered an exotic event in the literature with only few case studies and case series. So the aim of this study is to assess the risk of GI malignancies following primary GI carcinoids.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with gastrointestinal carcinoid tumor.
* patients diagnosed from 2000 till 2022

Exclusion Criteria:

* patients diagnosed with autopsy only or death certificate only.
* patients lacking age documentation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with gastrointestinal carcinoid tumor
Sampling Method: Probability Sample
Enrollment: 93481 (Actual)
Dates: Start 2000-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The standardized incidence ratio and excess risk of second primary gastrointestinal malignancies following primary gastrointestinal carcinoid tumors | Jan, 2000 till Dec, 2022
  The surveillance, epidemiology and End Results (SEER) database was used to calculate the standardized incidence ratio (SIR) as Observed/Expected (O/E) and calculated the excess risk for second primary gastrointestinal malignancies following primary gastrointestinal carcinoid tumors
The standardized incidence ratio and excess risk of gastrointestinal second primary malignancies stratified according to the primary gastrointestinal carcinoids site. | from Jan, 2000 till Dec, 2022

IPD SHARING:
Plan to Share IPD: Undecided